CLINICAL TRIAL: NCT00577564
Title: Endoscopic Ultrasound-guided Celiac Plexus Neurolysis (EUS-CPN): A Retrospective Review of Safety
Brief Title: EUS-CPN: A Retrospective Review
Status: Completed | Type: Observational
Sponsor: Indiana University (Other)
Responsible Party: Dr. Julia LeBlanc, Indiana University Medical Center
Other Study IDs: 0606-59; IRB #0606-59
Record Dates: First submitted 2007-12-19; First posted 2007-12-20 (Estimated); Last update posted 2012-09-12 (Estimated); Status verified 2012-09

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this retrospective study is to measure the safety of EUS-CPN in patients that have undergone this procedure in the last decade.

ELIGIBILITY:
Inclusion Criteria:

* Any subject that has undergone EUS-CPN will be considered for this study.

Exclusion Criteria:

* Subjects will be excluded if they have undergone a celiac plexus neurolysis (endoscopic, percutaneous, or surgical) at an another institution.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients that underwent a EUS-CPN over a ten year period at Indiana University Medical Center will be considered.
Sampling Method: Non-Probability Sample
Dates: Start 2006-07; Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Number of EUS-CPN procedures for each patient | over a ten year period

SECONDARY OUTCOMES:
Procedure-related complications | over a ten year period

CONTACTS AND LOCATIONS:
Overall Officials: Julia LeBlanc, MD, MPH, Principal Investigator — Indiana University School of Medicine
Locations (1):
- Clarian: University Hospital, Indianpolis, Indiana, United States